CLINICAL TRIAL: NCT03840369
Title: Pathophysiological Understanding and Treatment of PTSD: an rTMS Approach
Acronym: PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Defence Research and Development Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB18-1976
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-05

CONDITIONS: Stress Disorders, Post-Traumatic; Brain Injuries; Transcranial Magnetic Stimulation; Magnetic Resonance Spectroscopy; Biomarkers; Depression, Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Group 1: Treatment of the right dorsolateral prefrontal cortex Group 2: Treatment of the right dorsomedial prefrontal cortex
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS to the Right Dorsolateral Prefrontal Cortex (Experimental): Patients will engage in a one-week placebo control lead-in (5 treatments) and then a four-week treatment protocol (20 treatments) to the right Dorsolateral Prefrontal Cortex (DLPFC). The right DLPFC will be located with MR brain scans and the BrainSight TMS neuronavigation software. The intensity of the rTMS will be 100-120% of resting motor threshold amplitude, 1500 pulses applied consistently with a frequency of 1 Hz.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation to Right Dorsolateral Prefrontal Cortex; Device: Sham Repetitive Transcranial Magnetic Stimulation
- rTMS to the Right Dorsomedial Prefrontal Cortex (Experimental): Patients will engage in a one-week placebo control lead-in (5 treatments) and then a four-week treatment protocol (20 treatments) to the right Dorsomedial Prefrontal Cortex (DMPFC). The right DMPFC will be located with MR brain scans and the BrainSight TMS neuronavigation software. The intensity of the rTMS will be 100-120% of resting motor threshold amplitude, 1500 pulses applied consistently with a frequency of 1 Hz.
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation; Device: Repetitive Transcranial Magnetic Stimulation to Right Dorsomedial Prefrontal Cortex

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation to Right Dorsolateral Prefrontal Cortex — Transcranial magnetic stimulation (TMS) works by delivering a magnetic pulse to a focal brain region. TMS has a high degree of safety and has been studied as an intervention for many mental health and neurological conditions. Repetitive TMS (rTMS) delivers pulses at a set time interval in order to modulate neural activity in that region.
  Other Names: rTMS to DLPFC
  Arms: rTMS to the Right Dorsolateral Prefrontal Cortex
Device: Sham Repetitive Transcranial Magnetic Stimulation — The sham TMS coil will make a similar sound to the real rTMS coil, but will not deliver a magnetic pulse. This is a no-treatment device.
Device: Repetitive Transcranial Magnetic Stimulation to Right Dorsomedial Prefrontal Cortex — Transcranial magnetic stimulation (TMS) works by delivering a magnetic pulse to a focal brain region. TMS has a high degree of safety and has been studied as an intervention for many mental health and neurological conditions. Repetitive TMS (rTMS) delivers pulses at a set time interval in order to modulate neural activity in that region.
  Other Names: rTMS to DMPFC
  Arms: rTMS to the Right Dorsomedial Prefrontal Cortex

SUMMARY:
In Canada, the prevalence of PTSD is approximately 12%, similar to Canadian military personnel. Current treatments for PTSD are limited in efficacy and durability - indicating a dire need for novel interventions in this population. Transcranial magnetic stimulation (TMS) has a high degree of safety and has been studied as an intervention for many mental health and neurological conditions; even showing initial promise for PTSD. We propose to study this further in a randomized sham controlled trial of TMS for PTSD.

DETAILED DESCRIPTION:
In Canada, the prevalence of PTSD is approximately 12%, similar to Canadian military personnel. However, a 2002 study of members of Canadian Armed Forces found there was a striking positive correlation between the number of missions taken by the regular/reserve force and increase risk of developing PTSD, suggesting a dire need for further treatment options. Transcranial magnetic stimulation (TMS), a neuromodulation technique applied to the brain, has been studied as a treatment that has the potential to improve symptoms in a variety of neurological/mental health conditions. TMS is a safe and non-invasive technique that applies an electrical current to the brain to induce neuronal depolarization, changing regional brain function with the goal of improving neurological/psychiatric symptoms. Although multiple studies using TMS have suggested it as an efficacious treatment option for PTSD, clear knowledge gaps exist that prevent it from becoming evidence-based clinical care.

A recent meta-analysis on TMS and PTSD found that no study has examined the difference between genders, and recommended that further studies with larger sample sizes, equal male and female participants, and more stringent study designs were required. Our study is novel and seeks to bridge the gap from research to clinical care by completing a study investigating repetitive TMS (rTMS) treatment for PTSD that recruits a large sample size, uses a randomized controlled clinical trial with a sham lead-in, and follows a stringent TMS protocol with equal sex participants.

Not all individuals with PTSD respond to TMS treatment, and no study to date has explored what biomarkers may predict TMS responders in the PTSD population. Previous studies propose glutamate, BDNF and glutamatergic changes on MR spectroscopy may be altered in other mental health illnesses, which suggests they may be useful biomarkers of TMS response in PTSD. Therefore, this study will be the first of its kind to develop predictive biomarkers of response by sampling serum BDNF, glutamate, and glutamatergic changes in MR spectroscopy pre- and post rTMS treatment, in patients with PTSD that respond to TMS compared to those that do not.

Recent studies have shown single-pulse TMS is beneficial for some individuals with chronic PTSD, and emerging evidence suggests there are specific phenotypes within PTSD that may require different TMS protocols. A recent study by Etkin et al. explored whether there were multiple phenotypes within chronic PTSD that would explain treatment responses. They found individuals with PTSD that scored significantly lower on verbal memory tasks (LVMS) (list repetition) had significantly impaired functional connectivity in the brain's ventral attention network (VAN) compared to patients with PTSD that had normal scores (NVMS). This suggests there may be a subgroup of patients with PTSD that would respond better to TMS in the right dorsal medial prefrontal cortex (DMPFC) (corresponding to the VAN) than to the right dorsal lateral prefrontal cortex (DLPFC).

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants represent a typically developing nervous system as a more reliable target for this stage of research.
2. The presence of a PTSD diagnosis made by a physician will ensure participants are experiencing significant symptomatology and may benefit from treatment.
3. The cutoff score on the PCL-5 will ensure that participants are experiencing similar levels of symptoms to each other.
4. Need to have tried at least two types of treatment in the past

Exclusion Criteria:

1. Significant past medical history including seizures, stroke, severe traumatic brain injury, or central nervous system cancers may interfere with our evaluation of treatment outcome and will be criteria for exclusion.
2. Metal in head/neck/eye is a contraindication to safety in the MRI scanner and TMS protocol.
3. Women who are pregnant will not be included in the study due to potential risk of seizure during TMS. To determine if a patient is pregnant we will ask when their last menstrual cycle occurred. If there is a possibility of pregnancy, we will ask the participant to follow-up with their family doctor to confirm. We will then ask the participant to provide a written note from their treating practitioner stating they are not pregnant.
4. Active suicidality
5. Wellbutrin or benzodiazepine intake of more than 200mg/day, or more than 15 mg of Zopiclone per day as these medications lower seizure threshold
6. Trauma experienced less than a year ago and/or trauma experienced only as a child
7. Drug and/or alcohol abuse within the last 3 months (diagnosed by Canadian guidelines)
8. Diagnosed schizophrenia, untreated bipolar disorder, or psychosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Effect of 20-session rTMS Intervention to the DMPFC versus DLPFC on PCL Overall Score, Stratified by Verbal Memory Task Scores | Change in PCL-5 score at pre-treatment appointment, compared with the score at 1 week, upon study completion, and 4 weeks post-rTMS treatment.
  To determine whether patients with PTSD_LVMS have a greater response to a 20-day low frequency rTMS treatment protocol of the right DMPFC compared to the DLPFC, and if patients with PTSD_NVMS respond better to a 20-day low frequency TMS treatment protocol of the right DLPFC compared to the DMPFC as measured by the clinician administered PTSD scale for DSM-5 (CAPS-5) in male and female participants (military personnel and civilians) at 4 weeks and 1 month post-treatment.

SECONDARY OUTCOMES:
Serum BDNF, Glutamate, Glutathione, and MR Spectroscopy pre and post rTMS intervention | Change in serum BDNF, glutamate, and glutathione at the pre-treatment appointment compared with 1 week into treatment and upon study completion.
  To determine if serum brain derived neurotrophic factor (BDNF), glutamate, glutathione, and MR spectroscopy imaging will predict rTMS response in individuals with PTSD compared to those that do not respond to rTMS treatment.

OTHER OUTCOMES:
Effect of rTMS on Quality of Life After Brain Injury survey (QOLIBRI), headaches, anxiety and depression in individuals with PTSD | Change in QOLIBRI score at the pre-treatment appointment compared with 1 week, upon study completion, and 4 weeks post treatment.
  To determine if quality of life (QOLIBRI), including headaches, anxiety, and depression also improve with the rTMS treatment in individuals suffering with PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Foothill Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pohar R, Farrah K. Repetitive Transcranial Magnetic Stimulation for Patients with Depression: A Review of Clinical Effectiveness, Cost-Effectiveness and Guidelines - An Update [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Jun 28. Available from http://www.ncbi.nlm.nih.gov/books/NBK545105/ PMID 31433608
- [Background] Kobayashi M, Pascual-Leone A. Transcranial magnetic stimulation in neurology. Lancet Neurol. 2003 Mar;2(3):145-56. doi: 10.1016/s1474-4422(03)00321-1. PMID 12849236
- [Background] Vucic S, Kiernan MC. Transcranial Magnetic Stimulation for the Assessment of Neurodegenerative Disease. Neurotherapeutics. 2017 Jan;14(1):91-106. doi: 10.1007/s13311-016-0487-6. PMID 27830492
- [Background] Enokibara M, Trevizol A, Shiozawa P, Cordeiro Q. Establishing an effective TMS protocol for craving in substance addiction: Is it possible? Am J Addict. 2016 Jan;25(1):28-30. doi: 10.1111/ajad.12309. Epub 2015 Dec 21. PMID 26692110
- [Background] Lee JC, Blumberger DM, Fitzgerald PB, Daskalakis ZJ, Levinson AJ. The role of transcranial magnetic stimulation in treatment-resistant depression: a review. Curr Pharm Des. 2012;18(36):5846-52. doi: 10.2174/138161212803523644. PMID 22681165
- [Background] Kozel FA, Motes MA, Didehbani N, DeLaRosa B, Bass C, Schraufnagel CD, Jones P, Morgan CR, Spence JS, Kraut MA, Hart J Jr. Repetitive TMS to augment cognitive processing therapy in combat veterans of recent conflicts with PTSD: A randomized clinical trial. J Affect Disord. 2018 Mar 15;229:506-514. doi: 10.1016/j.jad.2017.12.046. Epub 2017 Dec 28. PMID 29351885
- [Background] Yan T, Xie Q, Zheng Z, Zou K, Wang L. Different frequency repetitive transcranial magnetic stimulation (rTMS) for posttraumatic stress disorder (PTSD): A systematic review and meta-analysis. J Psychiatr Res. 2017 Jun;89:125-135. doi: 10.1016/j.jpsychires.2017.02.021. Epub 2017 Feb 27. PMID 28278422
- [Background] Fryml LD, Sahlem G, Fox J, Short EB. The role of rTMS for patients with severe PTSD and depression. Evid Based Ment Health. 2018 Feb;21(1):39-40. doi: 10.1136/eb-2017-102819. Epub 2018 Jan 5. No abstract available. PMID 29305359
- [Background] Osuch EA, Benson BE, Luckenbaugh DA, Geraci M, Post RM, McCann U. Repetitive TMS combined with exposure therapy for PTSD: a preliminary study. J Anxiety Disord. 2009 Jan;23(1):54-9. doi: 10.1016/j.janxdis.2008.03.015. Epub 2008 Mar 28. PMID 18455908
- [Background] Wang HN, Bai YH, Chen YC, Zhang RG, Wang HH, Zhang YH, Gan JL, Peng ZW, Tan QR. Repetitive transcranial magnetic stimulation ameliorates anxiety-like behavior and impaired sensorimotor gating in a rat model of post-traumatic stress disorder. PLoS One. 2015 Feb 6;10(2):e0117189. doi: 10.1371/journal.pone.0117189. eCollection 2015. PMID 25659132
- [Background] Philip NS, Ridout SJ, Albright SE, Sanchez G, Carpenter LL. 5-Hz Transcranial Magnetic Stimulation for Comorbid Posttraumatic Stress Disorder and Major Depression. J Trauma Stress. 2016 Feb;29(1):93-6. doi: 10.1002/jts.22065. Epub 2016 Jan 7. PMID 26748883
- [Background] Pradhan B, Kluewer D'Amico J, Makani R, Parikh T. Nonconventional interventions for chronic post-traumatic stress disorder: Ketamine, repetitive trans-cranial magnetic stimulation (rTMS), and alternative approaches. J Trauma Dissociation. 2016;17(1):35-54. doi: 10.1080/15299732.2015.1046101. Epub 2015 Jul 10. PMID 26162001
- [Background] Watts BV, Landon B, Groft A, Young-Xu Y. A sham controlled study of repetitive transcranial magnetic stimulation for posttraumatic stress disorder. Brain Stimul. 2012 Jan;5(1):38-43. doi: 10.1016/j.brs.2011.02.002. Epub 2011 Mar 3. PMID 22264669
- [Background] Nam DH, Pae CU, Chae JH. Low-frequency, Repetitive Transcranial Magnetic Stimulation for the Treatment of Patients with Posttraumatic Stress Disorder: a Double-blind, Sham-controlled Study. Clin Psychopharmacol Neurosci. 2013 Aug;11(2):96-102. doi: 10.9758/cpn.2013.11.2.96. Epub 2013 Aug 26. PMID 24023554
- [Background] Oznur T, Akarsu S, Celik C, Bolu A, Ozdemir B, Akcay BD, Ozselek S, Bozkurt A, Ozmenler KN. Is transcranial magnetic stimulation effective in treatment-resistant combat related posttraumatic stress disorder? Neurosciences (Riyadh). 2014 Jan;19(1):29-32. PMID 24419446
- [Background] Berlim MT, Van Den Eynde F. Repetitive transcranial magnetic stimulation over the dorsolateral prefrontal cortex for treating posttraumatic stress disorder: an exploratory meta-analysis of randomized, double-blind and sham-controlled trials. Can J Psychiatry. 2014 Sep;59(9):487-96. doi: 10.1177/070674371405900905. PMID 25565694
- [Background] Novakovic V, Sher L, Lapidus KA, Mindes J, A Golier J, Yehuda R. Brain stimulation in posttraumatic stress disorder. Eur J Psychotraumatol. 2011;2. doi: 10.3402/ejpt.v2i0.5609. Epub 2011 Oct 17. PMID 22893803
- [Background] Liu G, Feng D, Wang J, Zhang H, Peng Z, Cai M, Yang J, Zhang R, Wang H, Wu S, Tan Q. rTMS Ameliorates PTSD Symptoms in Rats by Enhancing Glutamate Transmission and Synaptic Plasticity in the ACC via the PTEN/Akt Signalling Pathway. Mol Neurobiol. 2018 May;55(5):3946-3958. doi: 10.1007/s12035-017-0602-7. Epub 2017 May 26. PMID 28550530
- [Background] Moshe H, Gal R, Barnea-Ygael N, Gulevsky T, Alyagon U, Zangen A. Prelimbic Stimulation Ameliorates Depressive-Like Behaviors and Increases Regional BDNF Expression in a Novel Drug-Resistant Animal Model of Depression. Brain Stimul. 2016 Mar-Apr;9(2):243-50. doi: 10.1016/j.brs.2015.10.009. Epub 2015 Nov 10. PMID 26655599
- [Background] Hendrikse J, Kandola A, Coxon J, Rogasch N, Yucel M. Combining aerobic exercise and repetitive transcranial magnetic stimulation to improve brain function in health and disease. Neurosci Biobehav Rev. 2017 Dec;83:11-20. doi: 10.1016/j.neubiorev.2017.09.023. Epub 2017 Sep 23. PMID 28951250
- [Background] Lewis CP, Port JD, Frye MA, Vande Voort JL, Ameis SH, Husain MM, Daskalakis ZJ, Croarkin PE. An Exploratory Study of Spectroscopic Glutamatergic Correlates of Cortical Excitability in Depressed Adolescents. Front Neural Circuits. 2016 Nov 29;10:98. doi: 10.3389/fncir.2016.00098. eCollection 2016. PMID 27965544
- [Background] Etkin A, Maron-Katz A, Wu W, Fonzo GA, Huemer J, Vertes PE, Patenaude B, Richiardi J, Goodkind MS, Keller CJ, Ramos-Cejudo J, Zaiko YV, Peng KK, Shpigel E, Longwell P, Toll RT, Thompson A, Zack S, Gonzalez B, Edelstein R, Chen J, Akingbade I, Weiss E, Hart R, Mann S, Durkin K, Baete SH, Boada FE, Genfi A, Autea J, Newman J, Oathes DJ, Lindley SE, Abu-Amara D, Arnow BA, Crossley N, Hallmayer J, Fossati S, Rothbaum BO, Marmar CR, Bullmore ET, O'Hara R. Using fMRI connectivity to define a treatment-resistant form of post-traumatic stress disorder. Sci Transl Med. 2019 Apr 3;11(486):eaal3236. doi: 10.1126/scitranslmed.aal3236. PMID 30944165
- [Background] Kalita J, Laskar S, Bhoi SK, Misra UK. Efficacy of single versus three sessions of high rate repetitive transcranial magnetic stimulation in chronic migraine and tension-type headache. J Neurol. 2016 Nov;263(11):2238-2246. doi: 10.1007/s00415-016-8257-2. Epub 2016 Aug 19. PMID 27541044
- [Background] Cirillo P, Gold AK, Nardi AE, Ornelas AC, Nierenberg AA, Camprodon J, Kinrys G. Transcranial magnetic stimulation in anxiety and trauma-related disorders: A systematic review and meta-analysis. Brain Behav. 2019 Jun;9(6):e01284. doi: 10.1002/brb3.1284. Epub 2019 May 7. PMID 31066227
- [Background] Kozel FA. Clinical Repetitive Transcranial Magnetic Stimulation for Posttraumatic Stress Disorder, Generalized Anxiety Disorder, and Bipolar Disorder. Psychiatr Clin North Am. 2018 Sep;41(3):433-446. doi: 10.1016/j.psc.2018.04.007. PMID 30098656
- See also: National Center for PTSD — http://www.ptsd.va.gov/